CLINICAL TRIAL: NCT05924516
Title: Randomized Clinical Trial to Evaluate the Efficacy of a Digital Intervention for Patients With Type 2 Diabetes.
Acronym: DIAVERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria del Carmen Gogeascoechea Trejo (Other)
Collaborators: Adhera Health, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Maria del Carmen Gogeascoechea Trejo, PhD on Sciences Health, Universidad Veracruzana
Organization: Universidad Veracruzana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1284-0047
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Digital Interventions, mHealth, fatigue, behavioral
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatigue; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in two groups: control and experimental. Participants in the control group will continue with standard treatment, meanwhile participants in the experimental group will continue with standard treatment and will be enrolled in the digital intervention for 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control Group: Standard Treatment
- Experimental Group (Experimental): Experimental Group: Standard Treatment + Adhera® Fatigue Digital Program
  Interventions: Behavioral: Adhera® Fatigue Digital Program

INTERVENTIONS:
Behavioral: Adhera® Fatigue Digital Program — The Adhera® Fatigue Digital Program is delivered via a mobile application and includes personalized educational and interactive content. The program is designed to support the wellbeing of people living with type 2 diabetes, including self-management education and support. This also includes a focus on diabetes-related fatigue.
  Arms: Experimental Group

SUMMARY:
This study aims to perform a digital intervention in patients with type 2 diabetes to analyze the efficacy of the digital intervention Adhera® Fatigue Digital Program in order to improve diabetes self-management and improve clinical outcomes, including chronic condition-related fatigue. This will be done through a randomized clinical trial in 3 of the main health centers in the city of Xalapa, Veracruz, Mexico.

The digital health intervention is designed to be used for approximately 3 months. The study will enroll 150 participants (75 in control group and 75 in experimental group) who are patients with type 2 diabetes. There will be educational contents and personalized motivational messages through the Adhera Health Recommender System.

DETAILED DESCRIPTION:
Adhera® Fatigue Digital Program (or AFDP) T2D adaptation is a digital health program based on behavioral and emotional change techniques that provides support to patients with type 2 diabetes mellitus. The digital health solution is designed to be used for a period of 3 months and includes a mobile application that provides educational content and sends messages about 10 diabetes mellitus care areas with the aim of improving the quality of life of patients and therefore avoiding the occurrence of complications associated with the disease.

This is a clinical trial with 75 participants in the experimental intervention group and 75 in the control group, which will be carried out in 3 Primary Care Health centers in the City of Xalapa Veracruz, called Marabroto Center, Revolution Center and Miguel Alemán Center.

The researchers will focus on evaluating the main study variables to determine the changes in the indicators in glycosylated hemoglobin, total cholesterol, triglycerides, blood pressure, BMI, waist circumference and use of coping strategies.

The efficacy of the digital intervention will be measured in 2 ways: 1) Through the analysis of each of the study variables, where its decrease or increase represents that it was effective for the control of each indicator analyzed individually, and 2) Through the binary logistic regression model where all the variables of the study as a whole are analyzed and it is determined if the digital intervention had a global efficacy.

We believe that since it is a multifactorial disease, different variables that intervene in the complications of diabetes mellitus should be studied and not exclusively one single primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with type 2 diabetes mellitus diagnosed and treated in selected urban health centers of the Sanitary Jurisdiction V of Xalapa, Ver.
* Patients with smartphone and cell number.
* Participants must agree on sharing data from their clinical record.
* Participants must sign an informed consent.
* Participants must be willing to and install the mobile solution of the study.

Exclusion Criteria:

* Candidates without a smartphone or not being able to interact with it.
* Patients with type 1 diabetes mellitus, MODY (Maturity Onset Diabetes of the Young) and gestational diabetes.
* Patients who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (Hb1Ac) | Baseline
  The parameter will be measured in % reported in the control cards of the Health Centers where a normal level is <5.7%, prediabetes is between 5.7% to 6.4% and diabetes is above 6.5%. In patients with DM, 6 to 7% is a desired level, 7.1 to 8.5% is a moderate risk, 8.5 to 10% is a high risk, and 10% or more is a very high risk for the appearance of complications (WHO, 2021). This parameter will be retrieved from the site's health record of the study participants.
Glycosylated hemoglobin (Hb1Ac) | Month 3
  The parameter will be measured in % reported in the control cards of the Health Centers where a normal level is <5.7%, prediabetes is between 5.7% to 6.4% and diabetes is above 6.5%. In patients with DM, 6 to 7% is a desired level, 7.1 to 8.5% is a moderate risk, 8.5 to 10% is a high risk, and 10% or more is a very high risk for the appearance of complications (WHO, 2021). This parameter will be retrieved from the site's health record of the study participants.
Triglycerides | Baseline
  Triglycerides will be measured as an indicator of fat metabolism based on the fatty acid count (GPC, 2018). Its values are classified as normal <150 mg/dL; high limit of 150 to 199 mg/dL; high from 200 to 499 m/dL and very high 500 mg/dL and more. This parameter will be retrieved from the site's health record of the study participants.
Triglycerides | Month 3
  Triglycerides will be measured as an indicator of fat metabolism based on the fatty acid count (GPC, 2018). Its values are classified as normal <150 mg/dL; high limit of 150 to 199 mg/dL; high from 200 to 499 m/dL and very high 500 mg/dL and more. This parameter will be retrieved from the site's health record of the study participants.
Total Cholesterol | Baseline
  Total cholesterol, which includes lipoproteins of different density in the body, will be assessed (GPC, 2018). Its values are classified as normal when they are <200 mg/dL; intermediate high when they are between 200 and 239 mg/dL and high when they are above 240 mg/dL. This parameter will be retrieved from the site's health record of the study participants.
Total Cholesterol | Month 3
  Total cholesterol, which includes lipoproteins of different density in the body, will be assessed (GPC, 2018). Its values are classified as normal when they are <200 mg/dL; intermediate high when they are between 200 and 239 mg/dL and high when they are above 240 mg/dL. This parameter will be retrieved from the site's health record of the study participants.
Body Mass Index | Baseline
  It will be measured on the scale proposed by the WHO with the formula weight (kg) / height2 (mts) with the following categories: underweight <18.5; normal weight of 18.5-24.9; overweight: 24.9-29.9 and obesity >30. This parameter will be retrieved from the site's health record of the study participants.
Body Mass Index | Month 3
  It will be measured on the scale proposed by the WHO with the formula weight (kg) / height2 (mts) with the following categories: underweight <18.5; normal weight of 18.5-24.9; overweight: 24.9-29.9 and obesity >30. This parameter will be retrieved from the site's health record of the study participants.
Blood Pressure | Baseline
  It is classified as optimal <120/80 mmHg; normal 120-129/80-84 mmHg; high normal 130-139 mmHg/85-89 mmHg; grade 1 hypertension of 140-159/90-99 mmHg; grade 2 hypertension of 160-179/100-109 mmHg and grade 3 hypertension >180/>110 mmHg (WHO, 2021). This parameter will be retrieved from the site's health record of the study participants.
Blood Pressure | Month 3
  It is classified as optimal <120/80 mmHg; normal 120-129/80-84 mmHg; high normal 130-139 mmHg/85-89 mmHg; grade 1 hypertension of 140-159/90-99 mmHg; grade 2 hypertension of 160-179/100-109 mmHg and grade 3 hypertension >180/>110 mmHg (WHO, 2021). This parameter will be retrieved from the site's health record of the study participants.
Abdominal Perimeter | Baseline
  According to the CPG (2018) in men, an abdominal circumference <95 cm is considered normal, from 95 to 102 cm as a high risk for complications and >102 cm is considered a very high level of risk, while in women <82 cm is considered normal, 82 to 88 cm represents a high risk and <88 cm is a very high risk. This parameter will be retrieved from the site's health record of the study participants.
Abdominal Perimeter | Month 3
  According to the CPG (2018), in men an abdominal circumference <95 cm is considered normal, from 95 to 102 cm as a high risk for complications and >102 cm is considered a very high level of risk, while in women <82 cm is considered normal, 82 to 88 cm represents a high risk and <88 cm is a very high risk. This parameter will be retrieved from the site's health record of the study participants.
Use of coping strategies | Baseline
  It is based on the instrument "Coping Strategies Inventory (CSI)" prepared by Tobin et al., (1989) adapted by Cano et al., (2007) with a global evaluation of 0 to 160 points where the higher the score, the greater the use of coping strategies.
Use of coping strategies | Month 3
  It is based on the instrument "Coping Strategies Inventory (CSI)" prepared by Tobin et al., (1989) adapted by Cano et al., (2007) with a global evaluation of 0 to 160 points where the higher the score, the greater the use of coping strategies.

SECONDARY OUTCOMES:
Use of health services | Baseline
  The instrument to assess the use of health services during the last 3 months is entitled "Questionnaire on the use of health services attributable to diabetes mellitus" from Betz Brown et al., (2014) and does not have a representative scale, it only provides the number of times you have attended emergency services in the last 90 days. Ideally, a patient with DM under control should not go to the emergency or hospitalization services.
Use of health services | Month 3
  The instrument to assess the use of health services during the last 3 months is entitled "Questionnaire on the use of health services attributable to diabetes mellitus" from Betz Brown et al., (2014) and does not have a representative scale, it only provides the number of times you have attended emergency services in the last 90 days. Ideally in a patient with DM under control should not go to the emergency or hospitalization services.
Usability | Month 3
  It explores the degree to which a user evaluates the characteristics of the intervention, such as ease of use, simplicity, efficiency, information and user interface. It is supported by the Computer System Usability Questionnaire (CSUQ) from Hedlefs et al., (2016) and is classified as <28 points is deficient; 29-56 points is acceptable; 57-84 points is good and 85-112 points is favorable.

OTHER OUTCOMES:
Energy level | From week 1 to week 12, every two days
  It is measured on a scale from 1 to 10. It can be classified as low from 1 to 4, normal from 5 to 7, and high when the user values it from 8 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: María del Carmen Gogeascoechea Trejo, PhD, Study Director — Universidad Veracruzana
Locations (3):
- Mexico (3):
  - Clínic "José A. Maraboto" Street Santiago Bonilla 85, Xalapa, Veracruz
  - Clinic "Revolución" Street Valentín Canalizó, 12, Xalapa, Veracruz
  - Clinic "Miguel Alemán" Avenue Miguel Alemán 107, Xalapa, Veracruz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim EK, Kwak SH, Jung HS, Koo BK, Moon MK, Lim S, Jang HC, Park KS, Cho YM. The Effect of a Smartphone-Based, Patient-Centered Diabetes Care System in Patients With Type 2 Diabetes: A Randomized, Controlled Trial for 24 Weeks. Diabetes Care. 2019 Jan;42(1):3-9. doi: 10.2337/dc17-2197. Epub 2018 Oct 30. PMID 30377185
- [Background] Carrasco-Hernandez L, Jodar-Sanchez F, Nunez-Benjumea F, Moreno Conde J, Mesa Gonzalez M, Civit-Balcells A, Hors-Fraile S, Parra-Calderon CL, Bamidis PD, Ortega-Ruiz F. A Mobile Health Solution Complementing Psychopharmacology-Supported Smoking Cessation: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 27;8(4):e17530. doi: 10.2196/17530. PMID 32338624
- [Background] Brown JB, Ramaiya K, Besancon S, Rheeder P, Tassou CM, Mbanya JC, Kissimova-Skarbek K, Njenga EW, Muchemi EW, Wanjiru HK, Schneider E. Use of medical services and medicines attributable to diabetes in Sub-Saharan Africa. PLoS One. 2014 Sep 12;9(9):e106716. doi: 10.1371/journal.pone.0106716. eCollection 2014. PMID 25216268
- [Background] Cano Garcia FJ, Rodriguez Franco L, Garcia Martinez J. Spanish version of the Coping Strategies Inventory. Actas Esp Psiquiatr. 2007 Jan-Feb;35(1):29-39. PMID 17323223